CLINICAL TRIAL: NCT06045741
Title: Virtual Reality - A New Vision on Pain
Acronym: VROP
Status: Completed | Type: Observational
Sponsor: Sykehuset i Vestfold HF (Other)
Responsible Party: Principal Investigator, Inge Ringheim, PhD, Sykehuset i Vestfold HF
Other Study IDs: 21/00032
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pain; Pain, Chronic; Musculoskeletal Disorder; Musculoskeletal Pain; Musculoskeletal Diseases or Conditions; Musculoskeletal Neck Pain; Back Pain
Keywords: Virtual Reality; VR; Long lasting pain; Long-term
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Diseases; Musculoskeletal Pain; Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the project is to investigate if the use of virtual reality (VR) technology with pre-programmed proprietary software can provide better treatment for patients with long-term pain conditions. This is investigated in this pilot study conducted on patients referred to outpatient treatment at the Division of Physical Medicine and Rehabilitation. The pilot study will lay the foundation for a follow-up study (RCT). The effect of VR are evaluated by patient reporting forms; before start-up and 3 months after startup. Patients included in the study receive standard treatment supplemented with the use of VR technology.

The therapists involved will be Interviewed to examine their experiences with the use of the VR-technology in the treatment of patients.

VR technology can potentially contribute to better treatment (e.g. measured in outcomes such as activity, sleep problems, pain intensity, quality of life). Moreover we expect that a VR-assisted treatment to be more cost-effective and increased availability regardless of geography and demography.

ELIGIBILITY:
Inclusion Criteria:

* pain duration > 3 moths
* Master Norwegian spoken language

Exclusion Criteria:

* History of malignant disease
* pain duration < 3 Months
* Does not master Norwegian spoken language
* Epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain conditions, referred to the outpatient clinic at the division of physical medicine and rehabilitation at Vestfold Hospital Trust.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-08-18 (Actual); Study Completion 2024-08-18 (Actual)

PRIMARY OUTCOMES:
PROMIS Pain interference | Three months
  Consequences of pain on relevant aspects of one's life. This includes the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities.
  PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
PROMIS Pain intensity | Three months
  Numeric rating scale (NRS (0-10)) How much a person hurts

SECONDARY OUTCOMES:
System Usability Scale (SUS) | Three months
  The System Usability Scale (SUS) provides a reliable tool for measuring the usability. It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree.
EQ-5D-5L | Three months
  Health related quality of life; The Health Utilities Index is a rating scale used to measure general health status and health-related quality of life.
  Range fra
PROMIS Physical Function | Three months
  Self-reported capability rather than actual performance of physical activities. PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
PROMIS Emotional Distress - Anxiety | Three months
  Fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart,dizziness).
  PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
PROMIS Emotional Distress - Depression | Three months
  Negative mood (sadness, guilt), views of self (self- criticism,worthlessness), and social cognition (loneliness, interpersonal alienation), as well as decreased positive affect and engagement (loss of interest, meaning, and purpose).
  PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
PROMIS Physical Health - Sleep Disturbance | Three months
  Perceptions of sleep quality, sleep depth, and restoration associated with sleep.
  PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
PROMIS Social Health - Ability to Participate in Social Roles and Activities | Three months
  Perceived ability to perform one's usual social roles and activities. PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
PROMIS Physical Health - Fatigue | Three months
  Range of symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles.
  PROMIS measures are scored on the T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population.
RTWSE-11 Return ti work self efficacy | Three months
  The return to work self efficacy (RTW-SE) score quantifies an individual's confidence in their ability to work fully and perform work tasks while suffering from chronic pain conditions.
  The score ranges between 1 and 6, higher scores are better.
  Threshold values identified in Norwegian samples:
  Scores from 3.7 and lower are considered low and are associated with a lower probability of return to work. Scores from 4.6 and above are considered to be high and are associated with a higher probability of return to work.

CONTACTS AND LOCATIONS:
Locations (1):
- Klinikk fysikalsk medisin og rehabilitering, Sykehuset i Vestfold, Tønsberg, Norway

IPD SHARING:
Plan to Share IPD: No